CLINICAL TRIAL: NCT01930357
Title: Immunogenicity and Safety of the Purified Vero Rabies Vaccine - Serum Free (VRVg) in Comparison With the Human Diploid Cell Vaccine, Imovax® Rabies in a Pre-exposure Prophylaxis Regimen in Healthy Children and Adolescents Aged 2 to 17 Years
Brief Title: Purified Vero Rabies Vaccine-Serum Free Compared to Human Diploid Cell Vaccine in a Pre-exposure Prophylaxis Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VRV06; U1111-1127-7340 (Other: WHO); PHRR130822-000107 (Registry Identifier: The Philippine Health Research Registry (PHRR))
Record Dates: First submitted 2013-08-22; First posted 2013-08-28 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Rabies
Keywords: Rabies; Purified Vero Rabies Vaccine - Serum Free (VRVg); Imovax® rabies; Human Diploid Cell Vaccine
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VRVg Group (Experimental): Participants will receive receive 3 vaccinations of Purified Vero Rabies Vaccine Serum Free (VRVg)
  Interventions: Biological: Purified Vero Rabies Vaccine Serum Free (VRVg)
- Imovax® Rabies Group (Active Comparator): Participants will receive receive 3 vaccinations of Human Diploid Cell Vaccine (HDCV), Imovax® Rabies
  Interventions: Biological: Imovax® Rabies: Human Diploid Cell Vaccine (HDCV),

INTERVENTIONS:
Biological: Purified Vero Rabies Vaccine Serum Free (VRVg) — 0.5 mL, Intramuscular (Day 0, Day 7 and Day 28).
  Arms: VRVg Group
Biological: Imovax® Rabies: Human Diploid Cell Vaccine (HDCV), — 0.5 mL, Intramuscular (Day 0, Day 7 and Day 28).
  Other Names: Imovax® Rabies
  Arms: Imovax® Rabies Group

SUMMARY:
The aim of the study is to document immunogenicity and safety of VRVg in a pre-exposure regimen in healthy children and adolescents aged 2 to 17 years.

Primary Objectives:

* To demonstrate that VRVg is non-inferior to Imovax® Rabies in terms of proportion of subjects achieving a rabies virus neutralizing antibody (RVNA) titer ≥ 0.5 international units (IU)/mL at D42, i.e. 14 days after the last vaccination.
* To describe if at least 99% of subjects achieve an RVNA titer ≥ 0.5 IU/mL at D42 with a lower bound of the 95% confidence interval (CI) of at least 97%, in the VRVg group.

Secondary Objectives:

* To assess the clinical safety of each vaccine after each vaccine injection when administered in a pre-exposure schedule.
* To describe the immune response induced by each vaccine 14 days after the last vaccination, i.e. at D42, and 6 months after the first vaccination
* To describe the geometric mean titer ratio between the two vaccine groups at D42, i.e. 14 days after the last vaccination.

DETAILED DESCRIPTION:
Participants will receive a total of three vaccinations, one each at Day 0, Day 7, and Day 28, respectively, and will be assessment for immune response to rabies vaccine before the first injection (baseline titer), at Day 42, and at Month 6.

Safety will be assessed in all participants up to 28 days after each injection. Serious adverse events and adverse events of special interest (AESIs) will be collected up to 6 months after the last injection.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 to 17 years on the day of inclusion
* Informed consent form has been signed and dated by the parent(s) (and subject, if applicable by local regulations), or another legally acceptable representative and by an independent witness, as applicable, and the assent form has been signed and dated by the subject (if applicable by the local Ethics Committee or country regulations)
* Subject and parent/legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination)
* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine in the 4 weeks following any trial vaccination
* Any previous vaccination against rabies (in pre- or post-exposure regimen) with either the trial vaccine or another vaccine
* Bite by a potentially rabid animal in the previous 6 months without post-exposure prophylaxis
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to a vaccine containing any of the same substances
* Self-reported thrombocytopenia, contraindicating intramuscular vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* History of Guillain-Barré syndrome.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 342 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number Subjects with rabies virus neutralizing antibody (RVNA) titer ≥ 0.5 IU/mL as measured by rapid fluorescent focus inhibition test (RFFIT) | Day 42
  Rabies virus neutralizing antibody will be measured by rapid fluorescent focus inhibition test (RFFIT)

SECONDARY OUTCOMES:
Number of Participants Reporting Solicited Injection Site Reactions, Solicited Systemic Reactions, Unsolicited Systemic Reactions, and Serious Adverse Events Occurring Throughout the Trial | Day 0 up to 6 months post vaccination
  Solicited injection site reactions: pain, erythema, and swelling. Solicited systemic reactions: fever (temperature), headache, malaise, and myalgia
Summary Individual RVNA titer ratio (Day 42/Day 0) following vaccination with either Purified Vero Rabies Vaccine Serum Free (VRVg) or Human Diploid Cell Vaccine, Imovax® Rabies | Day 0 and Day 42
  Rabies virus neutralizing antibody will be measured by rapid fluorescent focus inhibition test (RFFIT)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (2):
- Philippines (2):
  - City of Muntinlupa
  - Manila

REFERENCES:
- [Derived] Quiambao B, Montalban C, Minutello AM, Guinet-Morlot F, Moureau A, Petit C, Pichon S. Serum-free purified Vero rabies vaccine is safe and immunogenic in children: Results of a randomized phaseII pre-exposure prophylaxis regimen study. Vaccine. 2022 Aug 19;40(35):5170-5178. doi: 10.1016/j.vaccine.2022.06.061. Epub 2022 Jul 26. PMID 35906106
- See also: Related Info — http://www.sanofipasteur.com